CLINICAL TRIAL: NCT03083561
Title: A Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3337641 in Japanese and Caucasian Healthy Subjects
Brief Title: A Study of LY3337641 in Japanese and Caucasian Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16174; I8K-JE-JPDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3337641 Multiple Dose (Experimental): Multiple doses of 30 mg LY3337641 tablet administered orally every day for two weeks, with a two week follow-up period.
  Interventions: Drug: LY3337641
- Placebo Multiple Dose (Placebo Comparator): Multiple doses of placebo administered orally every day for two weeks, with a two week follow-up period.
  Interventions: Drug: Placebo
- LY3337641 Single Dose (Experimental): Single dose of 5 mg, 80 mg and 160 mg LY3337641 tablet administered orally, with a two week follow-up period.
  Interventions: Drug: LY3337641
- Placebo Single Dose (Placebo Comparator): Single dose of placebo administered orally, with a two week follow-up period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3337641 — Administered orally.
  Arms: LY3337641 Multiple Dose; LY3337641 Single Dose
Drug: Placebo — Administered orally.
  Arms: Placebo Multiple Dose; Placebo Single Dose

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3337641 in healthy Japanese and Caucasian participants. The study will also investigate how the body processes LY3337641 and the effect of LY3337641 on the body. The study will last up to 4 weeks for each participant. Screening may occur within 28 days prior to first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese or Caucasian
* Body mass index (BMI) 18.0 - 32.0 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or off-label use of a drug or device or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer, if known) should have passed
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study or affects or confounds the QTc analysis or have Fridericia-corrected QT interval (QTcF) >450 milliseconds (msec) for males and >470 msec for females
* Have had symptomatic herpes zoster within 3 months of screening
* Have active or latent tuberculosis (TB) based on a positive medical history, examination, and/or TB test results.
* Have received live vaccine(s) within 1 month of screening or intend to during the study
* Are immunocompromised
* Have a history of constipation or have had acute constipation within 3 weeks prior to admission

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- WCCT Global, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of multiple-doses (MD) in Cohort 1 and single-dose (SD) for Cohorts 2, 3, and 4.
Groups:
- Placebo SD: Participants received single oral dose of placebo tablet with a two week follow-up period.
- 5 mg LY3337641 SD: Participants received single oral dose of 5 mg LY3337641 tablet with a two week follow-up period.
- 80 mg LY3337641 SD: Participants received single oral dose of 80 mg LY3337641 tablet with a two week follow-up period.
- 160 mg LY3337641 SD: Participants received single oral dose of 160 mg LY3337641 tablet with a two week follow-up period.
- Placebo MD: Participants received multiple oral doses of placebo tablet once daily for two weeks with a two week follow-up period.
- 30 mg LY3337641 MD: Participants received multiple oral doses of 30 mg LY3337641 tablet once daily for two weeks with a two week follow-up period.
Period: Overall Study
Arm/Group | Placebo SD | 5 mg LY3337641 SD | 80 mg LY3337641 SD | 160 mg LY3337641 SD | Placebo MD | 30 mg LY3337641 MD
Started | 6 | 6 | 6 | 6 | 3 | 9
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 3 | 9
Completed | 6 | 6 | 6 | 6 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SD | 5 mg LY3337641 SD | 80 mg LY3337641 SD | 160 mg LY3337641 SD | Placebo MD | 30 mg LY3337641 MD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.5) | 44.5 (10.1) | 46.7 (11.6) | 45.5 (12.0) | 36.0 (8.9) | 40.8 (12.5) | 43.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 2 | 3 | 15
  Male | 4 | 4 | 4 | 2 | 1 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 2 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 3 | 3 | 2 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 1 | 3 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 6 | 6 | 3 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Clinically significant events were defined as serious adverse events (SAE). A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Up To 31 Days
Population: All participants who received at least one dose of LY3337641 or placebo, and have at least one post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SD | 5 mg LY3337641 SD | 80 mg LY3337641 SD | 160 mg LY3337641 SD | Placebo MD | 30 mg LY3337641 MD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 3 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of LY3337641
Description: Cmax of LY3337641 was evaluated.
Time Frame: MD: Day 1 pre-dose, 0.25,0.5,1,2,3,4,6,8,10,12 and 24 hours post-dose,Day 15 pre-dose,0.25,0.5,1,2,3,4,6,8,10,12,24,36,48,96,168,240 and 336 hours post-dose. SD: pre-dose, 0.25,0.5,1,2,3,4,6,8,10,12,24,36,48,168 and 336 hours post-dose
Population: All participants who received at least 1 dose of LY3337641 and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- 5mg LY3337641 SD: Participants received single oral dose of 5 mg LY3337641 tablet with a two week follow-up period.
- 30mg LY3337641 MD Day 1: Participants received multiple oral doses of 30 mg LY3337641 tablet on day 1.
- 80mg LY3337641 SD: Participants received single oral dose of 80 mg LY3337641 tablet with a two week follow-up period.
- 160mg LY3337641 SD: Participants received single oral dose of 160 mg LY3337641 tablet with a two week follow-up period.
- 30mg LY3337641 MD Day 15: Participants received multiple oral doses of 30 mg LY3337641 tablet once daily for two weeks from day 1 to day 15
Arm/Group | 5mg LY3337641 SD | 30mg LY3337641 MD Day 1 | 80mg LY3337641 SD | 160mg LY3337641 SD | 30mg LY3337641 MD Day 15
Number analyzed (Participants) | 6 | 9 | 6 | 6 | 9
nanogram per milliliter (ng/mL) | 11.5 (56) | 56.5 (44) | 186 (25) | 358 (37) | 65.8 (54)

3. Secondary Outcome: PK: Area Under the Serum Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) of LY3337641
Description: AUC from zero to 24-hour of LY3337641 was evaluated.
Time Frame: MD: Day 1 pre-dose, 0.25,0.5,1,2,3,4,6,8,10,12 and 24 hours post-dose,Day 15 pre-dose,0.25,0.5,1,2,3,4,6,8,10,12 and 24 hours post-dose. SD: pre-dose, 0.25,0.5,1,2,3,4,6,8,10,12 and 24 hours post-dose
Population: All participants who received at least one dose of LY3337641 and have evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | 5mg LY3337641 SD | 30mg LY3337641 MD Day 1 | 80mg LY3337641 SD | 160mg LY3337641 SD | 30mg LY3337641 MD Day 15
Number analyzed (Participants) | 6 | 9 | 6 | 6 | 9
nanogram*hour per milliliter (ng*hr/mL) | 84.8 (58) | 276 (59) | 1040 (26) | 2100 (47) | 368 (65)

4. Secondary Outcome: PK: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3337641
Description: AUC from zero to infinity of LY3337641 was evaluated. For 30mg LY3337641 MD Day 1, pharmacokinetic data up to 24-hour post-dose were used for pharmacokinetic parameters calculation.
Time Frame: as for outcome 2
Population: All participants who received at least one dose of LY3337641 and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 5mg LY3337641 SD | 30mg LY3337641 MD Day 1 | 80mg LY3337641 SD | 160mg LY3337641 SD | 30mg LY3337641 MD Day 15
Number analyzed (Participants) | 6 | 9 | 6 | 6 | 9
ng*hr/mL | 92.0 (62) | 283 (61) | 1060 (27) | 2150 (48) | 382 (68)

ADVERSE EVENTS:
Time Frame: Up To 31 Days
Description: All enrolled participants.
Arm/Group | Placebo SD | 5 mg LY3337641 SD | 80 mg LY3337641 SD | 160 mg LY3337641 SD | Placebo MD | 30 mg LY3337641 MD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 1/6 | 2/6 | 3/3 | 6/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SD (N=6) | 5 mg LY3337641 SD (N=6) | 80 mg LY3337641 SD (N=6) | 160 mg LY3337641 SD (N=6) | Placebo MD (N=3) | 30 mg LY3337641 MD (N=9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT03083561/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03083561/SAP_001.pdf